CLINICAL TRIAL: NCT02788071
Title: Effect of Fecal Microbiota Transplantation in Irritable Bowel Syndrome (IBS) - a Randomized, Double-blind Placebo Controlled Pilot Study
Brief Title: Effect of Fecal Microbiota Transplantation in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aleris-Hamlet Hospitaler København (Other)
Collaborators: Hvidovre University Hospital (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Alice Højer Christensen, MD, PhD, Aleris-Hamlet Hospitaler København
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-15016343
Record Dates: First submitted 2016-05-30; First posted 2016-06-02 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Fecal Microbiota Transplantation; Microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT capsules (Experimental): FMT capsules
  Interventions: Dietary Supplement: FMT capsules
- FMT placebo (Placebo Comparator): Placebo capsules
  Interventions: Dietary Supplement: FMT placebo

INTERVENTIONS:
Dietary Supplement: FMT capsules — 25 capsules per day for 12 days
  Arms: FMT capsules
Dietary Supplement: FMT placebo — 25 capsules per day for 12 days
  Arms: FMT placebo

SUMMARY:
The purpose of this study is to investigate if fecal microbiota transplantation (FMT) will result in improvement in clinical outcome in patients with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is the most commonly diagnosed gastrointestinal condition. IBS is associated with a high use of health-care costs and can substantially reduce quality of life and work productivity.

Several studies have demonstrated that the composition of the gut microbiota in IBS patients is different from healthy controls.

Fecal microbiota transplantation (FMT) could therefore be a treatment option for IBS patients by exchanging the microbiota of an IBS patient with the microbiota of a healthy donor.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled Rome III diagnostic criteria for IBS
* Moderate-severe disease activity (IBS-Symptom Severity Score ≥175)
* Able to read and speak Danish
* Normal colonoscopy at age ≥ 40 years (performed within 1 year) or blood in stool

Exclusion Criteria:

* Other chronic gastrointestinal disease
* Positive fecal sample with enteropathogenic microorganisms or Clostridium difficile
* Positive screening for HIV, Hepatitis B or HCV antibody
* Surgical interventions in the gastrointestinal region (except for appendectomy, hernia repair, cholecystectomy, and gynecological and urological procedures)
* Psychiatric disorder
* Fecal calprotectin ≥ 50 mg/kg
* Abuse of alcohol or drugs
* Medications other than birth control pills, hormone supplements, allergies and asthma agents, blood pressure and cholesterol lowering agents, proton pump inhibitors and non-prescription medicines
* Abnormal screening biochemistry
* Abnormal colonoscopy findings
* Pregnant, planned pregnancy or breastfeeding females
* Ingestion of probiotics or antibiotics < 8 weeks before the inclusion

Inclusion criteria for donors

* Age between 18-45 years
* Past and current healthy
* Normal weight (BMI between 18,5-24,9 kg/m2)
* Normal bowel movements (defined as 1-2 per day and type 3-4 at Bristol Stool Form Scale)
* No medication consumption

Exclusion criteria for donors

* Known or high risk of infectious diseases such as HIV, hepatitis A, B or C
* Positive stool sample for C. difficile toxin, parasites or other pathogens
* Antibiotic treatment in the past 6 months
* Abuse of alcohol or drugs
* Smoking
* Tattoo or body piercing within the last 6 months
* Allergy, asthma or eczema
* Family history of gastrointestinal diseases
* Participation in high-risk sexual behaviors
* Born by Caesarean section

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
symptoms score | 12 weeks
  Measured by the Irritable bowel syndrome - severity symptom score (IBS-SSS)

SECONDARY OUTCOMES:
Change in microbiota diversity | Day 4, 4 weeks, 12 weeks and 24 weeks
  Measured by DNA sequencing
Microbiota diversity IBS patients | Baseline
  Measured by DNA sequencing
Microbiota diversity in healthy donors | Baseline
  Measured by DNA sequencing. To compare with the recipients (IBS patients)
Change in Irritable Bowel Syndrome-Quality of Life (IBS-QOL) Questionnaire Scores | Baseline, 4 weeks, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice Højer Christensen, MD, PhD, Principal Investigator — Aleris-Hamlet Hospitaler København
Locations (1):
- Aleris Hamlet Hospitaler, København, Copenhagen, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Halkjaer SI, Christensen AH, Lo BZS, Browne PD, Gunther S, Hansen LH, Petersen AM. Faecal microbiota transplantation alters gut microbiota in patients with irritable bowel syndrome: results from a randomised, double-blind placebo-controlled study. Gut. 2018 Dec;67(12):2107-2115. doi: 10.1136/gutjnl-2018-316434. Epub 2018 Jul 6. PMID 29980607